CLINICAL TRIAL: NCT00357292
Title: Comparison of the Ocular Tolerance, the Safety and the Ocular Pharmacokinetics After One Drop of Three Different Concentrations of T1225 (0.5% - 1.0% - 1.5%) in 48 Healthy Volunteers
Brief Title: Ocular Tolerance, Safety and Ocular Pharmacokinetics After 1 Drop of T1225 0.5, 1.0, 1.5% in 48 Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LT1225-PI1-09/01(AS)
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Last update posted 2006-07-27 (Estimated); Status verified 2006-07

CONDITIONS: Eye Infections, Bacterial
MeSH Terms: conditions — Eye Infections, Bacterial | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin (T1225)

SUMMARY:
To compare the ocular tolerance, the safety and the ocular pharmacokinetics of 3 concentrations (0.5% - 1.0% - 1.5%) and the vehicle of T1225 after one drop instillation

DETAILED DESCRIPTION:
The aim of the present study was to compare the ocular tolerance, safety and the ocular pharmacokinetics after a single administration of T1225 eye drops (0.5%, 1.0%, or 1.5%) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged from 18 to 45 years old;
* Written informed consent;
* Healthy volunteers (without any ocular symptom);
* Normal ocular examination in both eyes (corrected visual acuity (VA) >= 6/10 - Slit lamp examination without clinical relevant abnormalities - Tear break-up time (BUT) ≥10 seconds - Lachrymal secretion in the Schirmer test >= 10 mm in 5 minutes - Lissamine green test total score < 4 +).

Exclusion Criteria:

* Ocular trauma, infection or inflammation within the last 3 months;
* Blepharitis;
* Conjunctival hyperaemia (score >= 2 +);
* Watering (score >= 2);
* Contact lenses;
* Ocular surgery, including LASIK and PRK, within the last 12 months;
* Topical ocular treatment within the last month;
* Systemic antibiotics within the last 7 days;
* Any medication during the study (except: Paracetamol and contraceptives).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2002-03; Study Completion 2002-04

PRIMARY OUTCOMES:
Ocular subjective symptoms
Ocular objective symptoms

SECONDARY OUTCOMES:
Ocular pharmacokinetic.
Ocular and systemic adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Khalid TABBARA, Professor, Principal Investigator — The Eye Center, Riyadh (Saudi Arabia)